CLINICAL TRIAL: NCT00158548
Title: Studies on Adding Artesunate to Existing Antimalarial Therapies With Chloroquine, Amodiaquine & Sulphadoxine-pyrimethamine in Pakistan
Brief Title: ACT With Chloroquine, Amodiaquine & Sulphadoxine-pyrimethamine in Pakistan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: World Health Organization (Other); HealthNet TPO (Other); United Nations High Commissioner for Refugees (Other); Malaria Control Program, Directorate of Malaria Control, Pakistan (Other)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ITDCVC98; ITDCVV98
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Malaria; Falciparum Malaria; Vivax Malaria
Keywords: Falciparum; Vivax; Treatment; Asia
MeSH Terms: conditions — Malaria; Malaria, Falciparum; Malaria, Vivax | interventions — Chloroquine; Amodiaquine; Primaquine; Artesunate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: SP, chloroquine, amodiaquine, primaquine, artesunate

SUMMARY:
Chloroquine resistant falciparum malaria in Pakistan is prevalent in every malarious area examined. Resistance to the favoured second-line treatment, sulphadoxine-pyrimethamine S/P is rising fast. To avert a repetition of the resistance catastrophe that occurred in SE Asia it is critical to preserve the effective life of SP by using it in combination with artesunate. Efficacy of ACT with artesunate in combination with chloroquine, SP or amodiaquine for treatment of malaria (falciparum or vivax) will be examined in malaria patients in Pakistan.

DETAILED DESCRIPTION:
The incidence of falciparum malaria in Pakistan has risen 6-fold over the last 15 years and chloroquine resistance is prevalent in every malarious area examined. Chloroquine's position as first line treatment must be reconsidered. Resistance to the favoured second-line treatment, sulphadoxine-pyrimethamine SP, is 10% and rising fast. It is critical to preserve the effective life of SP by using it in combination with a non-related fast-acting antimalarial such as artesunate (AS). It is conceivable that use of AS in combination with chloroquine itself might even recover the latter's effectiveness and restrain the selection of stronger levels of chloroquine resistance. To determine the tolerability and efficacy of AS combination therapy in the subcontinent, randomized controlled trials will be conducted by HealthNet International and government staff, with technical support from LSHTM, in Afghan refugee camps in Pakistan against the current therapies of chloroquine, amodiaquine and SP. Current policy is to use primaquine(PQ) as the gametocytocidal drug with CQ or SP. It is not clear whether this has any value in the face of high levels of CQ resistance. The efficacy of PQ in combination with CQ or SP will be examined in individual randomised trial in comparison with CQ or SP alone.

In the past, treatment of falciparum and vivax malaria was with chloroquine. With development of drug resistance treatment of the two species is diverging and this places higher priority on accurate differential diagnosis which cannot always be met at peripheral health posts. There may be advantage in harmonising treatment of the two species with ACT. Thus the current treatment for vivax, chloroquine, shall be compared with that of ACT with artesunate and SP, the likely ACT to be adopted for falciparum malaria.

Protocol design:

Randomised, single-blind, controlled trials comparing for falciparum malaria (1) artesunate (AS) and chloroquine (CQ), vs CQ alone, vs CQ and primaquine (PQ); (2) AS and sulphadoxine-pyrimethamine (SP), vs SP alone, vs SP and PQ; (3) AS and amodiaquine (AQ), vs AQ alone.

Randomised, single-blind, controlled trial comparing for vivax malaria: AS and sulphadoxine-pyrimethamine (SP), vs CQ alone.

Patients will be randomly assigned to one of the following treatment groups:

* CQ (day1,2,3) + placebo (day 1, 3) vs
* CQ (day 1,2,3) + PQ (day 1) + placebo (day 3) vs
* CQ (day 1,2,3) + PQ (day 3) + placebo (day 1) vs
* CQ (day 1,2,3) + AS (day 1) + placebo (day 3)
* S/P (day 1) + placebo (day 1) vs
* S/P (day 1) + AS (day 1) vs
* S/P (day 1) + PQ (day 1)
* AQ (day 1,2,3) + placebo (day 1,2,3) vs
* AQ (day 1,2,3) + AS (day 1,2,3)

To determine the viability and transmissibility of any gametocytes (and also to detect sub-patent gametocytaemias) still present after treatment it is also proposed to carry out mosquito feeding studies directly on patients on the 7th day after the start of combination therapy with either CQ, CQ+AS, CQ+PQ., SP, SP+AS, SP+PQ and to incubate any midgut infections to the oocyst stage. To determine the genetic consequences of any selection from the different drugs (i.e. CQ, AS, or PQ), the mosquito midgut infections would be preserved for further genetic studies in UK, as would blood samples taken from initial and recrudescent infections.

To improve our understanding of the genetic basis of drug resistance we will genotype parasites from blood samples of patients with treatment failure in this study. Blood samples of 20 patients from each arm of the study who had parasitological treatment failure will be selected randomly, together with midgut infections, and analysed for genetic markers of resistance to chloroquine and sulphadoxine/pyrimethamine. These will be compared with genotypes of pre-treatment infections.

ELIGIBILITY:
Inclusion Criteria:

* adults or children > 5 yrs
* weight > 5 kg
* monoinfection with P. falciparum or P. vivax
* history of recent fever
* consent from patient or parent.

Exclusion Criteria:

* patients with signs of severe malaria.

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2001-06; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Day 7 slide clearance rate (complete clearance of trophozoites) assessed by microscopists who are blind to treatment allocation.
Day 28 slide clearance rate without subsequent recrudescence.
Day 7 gametocyte prevalence.

SECONDARY OUTCOMES:
Day 14 gametocyte prevalence
Fever clearance time
cure rate (elimination of parasitaemia without recrudescence).
Rate and time of parasite clearance.
Rate of resolution of fever.
Proportion of gametocyte carriers.
Transmissibility of gametocytes through mosquito feeding studies.
Tolerability.
Molecular characterisation of genetic diversity and resistance before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Graham, MSc, Principal Investigator — HealthNet International, Peshawar, Pakistan
Locations (1):
- HealthNet International, Peshawar, Pakistan